CLINICAL TRIAL: NCT00238212
Title: Phase II Study of BAY 43-9006 (NSC #724772) as Single Agent in Unresectable or Metastatic Gallbladder Carcinoma and Cholangiocarcinoma
Brief Title: S0514 Sorafenib in Treating Patients With Unresectable or Metastatic Gallbladder Cancer or Cholangiocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03181; S0514; U01CA32102 (Other Grant/Funding Number: US NIH Grant/Contract Award Number); CDR0000444959 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Adenocarcinoma of the Extrahepatic Bile Duct; Adenocarcinoma of the Gallbladder; Adenocarcinoma With Squamous Metaplasia of the Gallbladder; Cholangiocarcinoma of the Extrahepatic Bile Duct; Cholangiocarcinoma of the Gallbladder; Recurrent Extrahepatic Bile Duct Cancer; Recurrent Gallbladder Cancer; Squamous Cell Carcinoma of the Gallbladder; Unresectable Extrahepatic Bile Duct Cancer; Unresectable Gallbladder Cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — Sorafenib

ARMS (1):
- Treatment (Experimental): Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well sorafenib works in treating patients with unresectable or metastatic gallbladder cancer or cholangiocarcinoma. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the objective response probability (complete responses and partial responses) for BAY 43-9006 in patients with unresectable or metastatic gallbladder or cholangiocarcinoma.

II. To assess overall survival, time to treatment failure and progression-free survival in these patients.

III. To assess quantitative and qualitative toxicities of this regimen. IV. To evaluate in a preliminary fashion relevant prognostic and predictive molecular markers of clinical outcome in gallbladder and cholangiocarcinoma.

OUTLINE: This is a multicenter study.

Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a cytologically or pathologically confirmed diagnosis of cholangiocarcinoma or gallbladder carcinoma

  * The pathologic confirmation of gallbladder or cholangiocarcinoma may be made from the primary or metastatic site; biopsy of the gallbladder or bile duct mass is not necessary; patients with pathologic confirmation of adenocarcinoma of a metastatic site, along with clinical documentation of gallbladder or bile duct involvement and no evidence of another primary are also eligible; if clinical documentation of gallbladder or bile duct involvement is not possible because of removal of the organ, a clinically and/or radiographically consistent picture plus pathologic findings from the metastatic site that are determined to be consistent with cholangiocarcinoma are acceptable
  * Eligible pathologic type: Patient must have one of the following subtypes: adenocarcinoma NOS, papillary carcinoma, adenocarcinoma, intestinal type, clear cell adenocarcinoma, mucinous adenocarcinoma, signet ring cell carcinoma, squamous cell carcinoma, adenosquamous carcinoma, small cell carcinoma, undifferentiated carcinoma, carcinoma NOS; patient must not have carcinoid tumors or sarcomas
* Patient must have locally advanced or distant metastatic disease that is not surgically curable
* Patient must have measurable disease; x-rays, scans or physical examinations used for tumor measurement must have been completed within 28 days prior to registration; x-rays, scans or other tests for assessment of non-measurable disease must have been performed within 42 days prior to registration; all disease must be assessed
* Institutions are required to submit paraffin-embedded specimens
* Institutions are required to seek additional patient consent for submission of blood
* Patient may have had prior surgery, including surgery for their gallbladder or cholangiocarcinoma; patients must be at least 14 days beyond any major surgery, and recovered from all effects of surgery
* Patient must not have received prior therapy for unresectable or metastatic disease; patient may have received prior chemotherapy, hormonal therapy, immunotherapy, radiation therapy (to less than 25% of bone marrow only) or chemoradiotherapy as neoadjuvant or adjuvant treatment; this must have been completed at least 12 months prior to documented recurrence or metastatic disease; patient must have recovered from all radiation induced toxicities
* Prior radiation therapy to metastatic sites, such as bone, is allowed as long as the patient has measurable lesion(s) that were not treated with radiation therapy; at least 28 days must have elapsed since completion of radiation therapy, and patient must have recovered from all effects
* Patient must not have received prior BAY 43-9006 or any inhibitor of VEGFR or the MAPK pathway
* Patient must have Zubrod performance status of 0-1
* Total serum bilirubin =< 3 x the institutional upper limit of normal (IULN)
* Serum transaminase (SGOT or SGPT) =< 2.5 x IULN; if liver metastasis is present, SGOT or SGPT must be =< 5 x IULN
* Patients with biliary obstruction must have decompressions of the biliary tree by ERCP and stenting or percutaneous drainage
* Serum creatinine =< 1.5 x IULN OR measured creatinine clearance >= 60 mL/min OR estimated creatinine clearance >= 60 mL/min
* Leukocyte count >= 3,000/mcL
* ANC >= 1,000/mcL
* Platelets >= 100,000/mcL
* PT, INR and PTT =< IULN
* Patients must not be taking the cytochrome P450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine, and Phenobarbital), rifampin, or St. Johns Wort
* Patient must not be on therapeutic anticoagulation; prophylactic anticoagulation (i.e., low dose warfarin) of venous or arterial access devices is allowed provided that the requirements for PT, INR and PTT are met
* Patient must not have any evidence of bleeding diathesis
* Patients must not have clinically significant cardiac disease that is not well controlled by medication (e.g., congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias) or myocardial infarction within 12 months prior to registration
* Patient must not have uncontrolled hypertension
* Patient must not have known brain metastases because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Patient must either be able to swallow and/or receive enteral medications via gastrostomy feeding tube; tablets must not be crushed; patient must have the ability to absorb medication (i.e., no malabsorption syndrome); patient must not have intractable nausea or vomiting
* Patient must have no plans to receive concurrent chemotherapy, hormonal therapy, radiotherapy, immunotherapy or any other type of therapy for treatment of cancer while on this protocol; radiation for palliation to metastatic sites is allowed as long gas the target lesions are not irradiated
* Women/men of reproductive potential must agree to use an adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of protocol treatment; post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential; pregnant or nursing women are not eligible for this protocol; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; breastfeeding must be discontinued if the mother is treated with BAY 43-9006
* HIV-positive patients must have a CD4 count > 500 and must have no active opportunistic infection; in addition, patient must not be receiving combination anti-retroviral therapy
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years
* If day 14, 28 or 42 falls on a weekend or holiday, the limit may be extended to the next working day

  * In calculating days of tests and measurements, the day a test or measurement is done is considered day 0; therefore, if a test is done on a Monday, the Monday two weeks later would be considered day 14; this allows for efficient patient scheduling without exceeding the guidelines
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and ID number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-10; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Response probability (confirmed complete and confirmed partial responses) | Up to 3 years

SECONDARY OUTCOMES:
Overall survival | From date of registration to date of death due to any cause, assessed up to 3 years
Time to treatment failure | From date of registration to date of first observation of progressive disease, death due to any cause, symptomatic deterioration, or early discontinuation of treatment, assessed up to 3 years
Time to progression | From date of registration to date of first observation of progressive disease, death due to any cause or symptomatic deterioration, assessed up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Anthony El-Khoueiry, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group, San Antonio, Texas, United States